CLINICAL TRIAL: NCT05740618
Title: Effect of Bronchitol on Mucociliary Clearance in Cystic Fibrosis Transmembrane Conductance Regulator (CFTR)-Modulator Treated Patients With Cystic Fibrosis With Moderate to Severe Lung Disease
Brief Title: Inhaled Mannitol on Mucociliary Clearance in Moderate to Severe Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Chiesi USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-1790
Record Dates: First submitted 2023-02-03; First posted 2023-02-23 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Inhaled Mannitol (Experimental): All study participants will receive the same study treatment. Study treatment will be dry powder mannitol 400 mg twice a day by oral inhalation (the contents of 10 capsules administered individually) for 14 days +/- 2 days.
  Interventions: Drug: Mannitol Inhalant Product

INTERVENTIONS:
Drug: Mannitol Inhalant Product — A sugar alcohol indicated as an add-on maintenance therapy to improve pulmonary function in adult patients 18 years of age and older with cystic fibrosis.
  Other Names: Bronchitol; dry powder mannitol

SUMMARY:
This study will provide important mechanistic information regarding the effect of inhaled mannitol (Bronchitol) in people with cystic fibrosis (PwCF) with moderate to severe disease who are already using elexacaftor/tezacaftor/ivacaftor (E/T/I). Many patients have already discontinued hypertonic saline and other pulmonary therapies because of the profound effect of E/T/I of their symptoms and lung function. Further, because both inhaled osmotic agents (i.e., Bronchitol, hypertonic saline [HS]) and E/T/I are believed to exert their beneficial effects through improvements in mucociliary clearance (MCC), it is unknown if the combination of these therapies might be additive or are redundant in a population with moderate to severe disease where bronchiectasis and chronic infection persists, and where eventual decline in lung function is expected over time. This study, therefore, will be the first to determine whether "add on" therapy with inhaled mannitol is able to further accelerate MCC in E/T/I patients. These data would provide some guidance regarding the use of these approved therapies in PwCF.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Age ≥ 18 at the time of screening
* Diagnosis of cystic fibrosis (CF)
* Regularly using elexacaftor/tezacaftor/ivacaftor (E/T/I) for ≥ 90 days
* Forced Expiratory Volume in one second (FEV1) between 30% and 70%, inclusive, at time of screening
* Denies active smoking or vaping
* Clinically stable with no significant changes in health status within the 28 days prior to and including the screening visit
* Patients on cycled inhaled antibiotics will need to be either on or off their antibiotic for 7 days prior to Visit 1 and not scheduled to cycle during the 2-week treatment period until after Visit 2
* Has no other conditions that, in the opinion of the Site Investigator/Designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Exclusion Criteria:

* Use of an investigational drug within 28 days prior to and including the screening visit
* Unable or unwilling to withhold hypertonic saline (HS) for 4 weeks (2 weeks prior to Visit 1 and 2 weeks between Visit 1 and Visit 2)
* Unable or willing to withhold dornase alfa and bronchodilators on the morning of Visit 1 and Visit 2, until completion of study procedures
* Initiation of new chronic CF pulmonary therapy (e.g. dornase alfa, azithromycin, inhaled antibiotic) within 28 days prior to and including the screening visit
* No acute use of antibiotics (oral, inhaled, or intravenous) or acute use of systemic corticosteroids for respiratory tract symptoms within 28 days prior to and including the screening visit.
* No chronic use of oral corticosteroids > 10 mg of prednisone or equivalent daily
* Unable to tolerate albuterol or other bronchodilator
* History of intolerance to HS or inhaled mannitol
* Pregnancy or breast feeding
* Have had more than 2 chest computed tomography (CT) in the past year or a combination of procedures that are believed to have exposed the subject's lungs to >150 millisievert (mSv)
* History of significant hemoptysis (>60 mL) in the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhashini A Sellers, MD, MSCR, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled Mannitol
Started | 14
Completed | 12
Not Completed | 2
Not completed — Did not meet Inclusion/Exclusion criteria | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Inhaled Mannitol
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Baseline Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: percent predicted] | 48.6 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Average Rate of Mucociliary Clearance (MCC) Over 60 Minutes
Description: A whole lung region of interest (ROI) bordering the right lung is used to estimate (by computer analysis) whole lung retention of inhaled radiolabeled particles. Labeled particle counts are measured over a 60-minute period to determine the fraction of initial particle counts remaining. From this data, the investigators will determine the percentage of labeled particles cleared from the lung during the 60-minute observation period. The primary outcome will be expressed as a percent, representing total average rate of mucociliary clearance (MCC) in the whole right lung compartment over 60 minutes (MCC60).
Time Frame: Day 14 (+/-2 days)
Measure: Mean (Standard Deviation); unit: percent cleared over 60 minutes
Arm/Group | Inhaled Mannitol
Number analyzed (Participants) | 12
percent cleared over 60 minutes | 14.8 (6.5)
Statistical Analysis 1: Comparison: Inhaled Mannitol; Test type: Superiority; p = 0.04, Mixed Models Analysis — MCC60 was analyzed using a linear repeated measure model including visit number, skew of the deposition histogram as fixed effects

2. Secondary Outcome: Cough Clearance
Description: Subjects will cough a total of 30 times over a 30-minute period to assess cough clearance by gamma imaging over that period. Clearance will be determined by measuring the decrease in radiolabeled Tc99m-sulfur colloid in the lungs over time expressed as a percent cleared.
Time Frame: Day 14 (+/-2 days)
Measure: Mean (Standard Deviation); unit: percent cleared over 30 minutes
Arm/Group | Inhaled Mannitol
Number analyzed (Participants) | 12
percent cleared over 30 minutes | 0.30 (0.06)
Statistical Analysis 1: Comparison: Inhaled Mannitol; Test type: Superiority; p = 0.20, t-test, 2 sided — T-tests performed as paired analyses using baseline cough clearance

3. Secondary Outcome: Rate of Mucociliary Clearance (MCC) Over 90 Minutes
Description: A whole lung region of interest (ROI) bordering the right lung is used to estimate (by computer analysis) whole lung retention of inhaled radiolabeled particles. Labeled particle counts are measured over a 90-minute period to determine the fraction of initial particle counts remaining. From this data, the investigators will determine the percentage of labeled particles cleared from the lung during the 90-minute observation period. The primary outcome will be expressed as a percent, representing total average rate of mucociliary clearance (MCC) in the whole right lung compartment over 90 minutes (MCC90).
Time Frame: Day 14(+/-2 days)
Measure: Mean (Standard Deviation); unit: percent cleared over 90 minutes
Arm/Group | Inhaled Mannitol
Number analyzed (Participants) | 12
percent cleared over 90 minutes | 18.2 (7.7)
Statistical Analysis 1: Comparison: Inhaled Mannitol; Test type: Superiority; p = 0.07, t-test, 2 sided — T-tests performed as paired analyses using baseline Mucociliary Clearance (MCC) Over 90 Minutes

4. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Percent of Predicted
Description: FEV1 is measured by spirometry. On each occasion, the best of 3 trials, based on American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria. The best FEV1 (from trial with highest sum of FEV1 and Forced Vital Capacity (FVC)) will be recorded and reported as percent of predicted.
Time Frame: Day 14 (+/-2 days)
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Inhaled Mannitol
Number analyzed (Participants) | 12
percent predicted | 46.9 (11.3)
Statistical Analysis 1: Comparison: Inhaled Mannitol; Test type: Superiority; p = 0.04, t-test, 2 sided — T-tests performed as paired analyses using baseline FEV1

5. Secondary Outcome: Respiratory Symptoms as Measured by the Cystic Fibrosis Respiratory Questionnaire Revised (CFQR-R)
Description: The CFQ-R (Cystic fibrosis Questionnaire - Revised) is a detailed, rigorously designed and validated self-report instrument designed to measure quality of life in patients with CF who are 14 years and older. This instrument was developed as the first CF-specific, health-related Quality of Life (QOL) measure. The respiratory domain has a 0-100 scale, with higher values signifying less severe symptoms.
Time Frame: Day 14(+/-2 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inhaled Mannitol
Number analyzed (Participants) | 12
score on a scale | 78.3 (13.7)
Statistical Analysis 1: Comparison: Inhaled Mannitol; Test type: Superiority; p = 0.94, t-test, 2 sided — T-tests performed as paired analyses using baseline CFQR-R respiratory domain

6. Secondary Outcome: Respiratory Symptoms as Measured by the Cystic Fibrosis Respiratory Symptom Diary and Chronic Respiratory Infection Symptom Score (CFRSD-CRISS)
Description: The CFRSD-CRISS is an 8-item, patient-centered, self-report outcome measure evaluating symptom severity over the prior 24 hours in 8 domains central to CF. Each question is assigned a score from 0-4 based on the response, with zero reflecting the absence of the symptom and four reflecting that the symptoms is present 'a great deal' or 'extremely'. A summed score (range from 0-24) is converted to a 0-100 scale, where lower scores indicate fewer symptoms.
Time Frame: Day 14(+/-2 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inhaled Mannitol
Number analyzed (Participants) | 12
score on a scale | 33.3 (7.2)
Statistical Analysis 1: Comparison: Inhaled Mannitol; Test type: Superiority; p = 0.13, t-test, 2 sided; T-tests performed as paired analyses using baseline CFRSD-CRISS

7. Secondary Outcome: Respiratory Symptoms as Measured by the Treatment Satisfaction Questionnaire Measure (TSQM)
Description: The TSQM is a 14-question standardize measure for assessment of self-reported treatment satisfaction and has been valued for use of inhaled medications in people with CF. The TSQM items are answered on 5- or 7-point Likert type scale and cover four domains, corresponding to distinct aspects related to the satisfaction of patients with their treatment (Effectiveness; Side effects; Convenience and Global satisfaction). The questionnaire is scored on a 0-100 scale, with higher values indicated greater satisfaction.
Time Frame: Day 14(+/-2 days)
Population: While participants completed the questionnaire, we are unable to generate a reportable result. As we learned late in the process, the scoring manual required to code responses and calculate results is proprietary, and the rights for its use were not secured. This data will never be analyzed in the future. The study protocol was not amended to reflect this change.
Arm/Group | Inhaled Mannitol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through Visit 2 completion, up to 4 weeks.
Arm/Group | Inhaled Mannitol
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Mannitol (N=13)
Inhaled mannitol intolerance as demonstrated by FEV1 decline (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT05740618/Prot_SAP_000.pdf